CLINICAL TRIAL: NCT05283356
Title: Single Antiplatelet Treatment With Ticagrelor or Aspirin After Transcatheter Aortic Valve Implantation: Multicenter Randomized Clinical Trial
Brief Title: Single Antiplatelet Treatment With Ticagrelor or Aspirin After Transcatheter Aortic Valve Implantation
Acronym: REAC-TAVI2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REAC-TAVI 2; 2021-003927-13 (EudraCT Number)
Record Dates: First submitted 2022-03-01; First posted 2022-03-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Severe Aortic Valve Stenosis; Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement (TAVR); Transcatheter Aortic Valve Implantation (TAVI)
Keywords: Severe Aortic Valve Stenosis; Transcatheter aortic valve replacement (TAVR); Transcatheter aortic valve implantation (TAVI); Single antiplatelet therapy (SAPT); Ticagrelor 60 mg; ASA 100 mg; Bleeding; Valve thrombosis
MeSH Terms: conditions — Aortic Valve Stenosis; Hemorrhage | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetylsalicylic acid 100mg/day (Active Comparator): Aspirin 100 mg/day after TAVI
  Interventions: Drug: Ticagrelor 60mg
- Ticagrelor 60mg twice per day (Experimental): Ticagrelor 60 mg twice per day after TAVI
  Interventions: Drug: Ticagrelor 60mg

INTERVENTIONS:
Drug: Ticagrelor 60mg — Ticagrelor 60mg BID after TAVI

SUMMARY:
The optimal pharmacological therapy after transcatheter aortic valve implantation (TAVI) to prevent valve thrombosis and reduce thromboembolic complications without significantly increasing the risk of bleeding is not yet fully defined and constitutes an important unmet clinical need. Recently, single antiplatelet therapy (SAPT) with Aspirin has been increasingly adopted to avoid bleeding early after TAVI compared with dual antiplatelet therapy. However, TAVI population is affected by a diversity of chronic pathologies that increase the risk of post-TAVI ischemic complications. Stroke is prevalent, especially peri- and early post-TAVI (<1-8% in the 1st year). Although peri-TAVI myocardial infarction (MI) is rare (1-3%), concomitant coronary artery disease (CAD), diabetes mellitus (DM), and peripheral vascular disease (PVD), is very frequent in the TAVI population, affecting around 30-70% of patients. In patients with CAD, the need to re-access the coronary arteries after TAVI is challenging and can be hampered by the trancatheter valve struts.

This is critical in TAVI patients with an acute coronary syndrome and in younger patients with long-life expectancy after TAVI. The use of a P2Y12 inhibitor provides significant ischemic protection in the in the coronary, cerebral and peripheral vascular territories compare to Aspirin. The use of a P2Y12 inhibitor as antiplatelet treatment can decrease the need for new coronary revascularizations and reduce the incidence of thromboembolic complications after TAVI.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Adult patients (more than 18 years) with ability to understand and accept the participation in the clinical trial.
3. Patients with degenerative symptomatic severe aortic stenosis (AS) accepted for TAVI with any of the commercial approved TAVI devices after evaluation of the Heart Team of each center,and with at least one of the following comorbidities:

   1. Diabetes Mellitus, the current WHO diagnostic criteria for diabetes should be maintained - fasting plasma glucose ≥ 7.0mmol/l (126 mg/dl) or 2-h plasma glucose ≥ 11.1mmol/l (200mg/dl), or under treatment with an oral hypoglycemic or insulin.
   2. Prior coronary artery disease (STEMI, NSTEMI, stable angina, or others) documented by invasive or non-invasive ischemia screening tests or imaging study.
   3. Prior peripheral arterial disease documented by invasive or non-invasive ischemia screening tests or imaging study.
4. Successful TAVI performed by any vascular access.
5. Patients who are not participating in any other clinical trial or research study (registries allowed).

Exclusion Criteria:

1. Patients under chronic oral anticoagulation for any specific pathology.
2. Patients that cannot undergo a regimen of single antiplatelet therapy after TAVI.
3. History of overt major bleeding or intracranial hemorrhage.
4. Active pathological bleeding.
5. History of ischemic stroke within the last 30 days prior TAVI.
6. Patients with documented severe hepatic insufficiency.
7. Known pregnancy, breast-feeding, or intend to become pregnant during the study period.
8. Concomitant oral or intravenous therapy with potent inhibitors of cytochrome P450 3A (CYP3A) that cannot be suspended during the study.
9. Patients randomized in another clinical trial with an investigational product or device over the past 30 days.
10. Patients who cannot attend follow-up visits scheduled in the study.
11. History of allergic reactions or intolerance to Ticagrelor or Aspirin or any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1206 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of Ticagrelor vs Aspirin in the incidence of NACE at 12 months after TAVI. | 12 months
  NACE is a composite of: all-cause mortality, transient ischemic attack (TIA) or stroke, myocardial infarction, progressive angina leading to emergency evaluation,rehospitalization or new coronary angiography, valve thrombosis, claudication, acute limb ischemia leading to hospitalization, any bleeding.

SECONDARY OUTCOMES:
Efficacy endpoint: Subclinical valve thrombosis | 3 and 12 months
  Detected by hypoattenuated leaflet thickening (HALT) and reduced leaflet motion(RLM) at 3 and 12 months after TAVI assessed by 4-dimensional computed tomography (4D-CT) imaging.
  HALT: Hypoattenuating thickening in typically meniscal configuration on one or more leaflets, with or without RLM. The extent of HALT should be described per leaflet, using a 4-tier grading scale in regard to leaflet involvement along the curvilinear contour, assuming maximum involvement at the base of the leaflet:
  ≤25% (limited to the base) >25% and ≤50% >50% and ≤75% >75% Inconclusive for HALT: imaging with insufficient image quality or presence of artifact RLM: The extent of RLM should be described per leaflet, using a 4-tier grading scale None: no reduction in leaflet excursion <50% reduction in leaflet excursion
  ≥50% reduction in leaflet excursion Immobile: immobile leaflet Inconclusive for RLM: imaging with insufficient image quality or presence of artefact
Safety endpoint: Major bleeding | 12 months
  Major bleeding (type 2, 3 and 5) at 12 months after TAVI according BARC (Bleeding Academic Research Consortium)
Patient-oriented composite endpoints | 12 months
  Patient-oriented composite endpoints (POCE) at 12 months after TAVI (POCE is a composite of all-cause mortality,TIA/stroke, myocardial infarction, progressive angina leading to emergency evaluation, rehospitalization or new coronary angiography).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Alvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jimenez Diaz VA, Lozano I, Tello Montoliu A, Baz Alonso JA, Iniguez Romo A. Is There a Link Between Stroke, Anticoagulation, and Platelet Reactivity?: The Multifactorial Stroke Mechanism Following TAVR. JACC Cardiovasc Interv. 2019 Dec 23;12(24):2560-2561. doi: 10.1016/j.jcin.2019.10.004. No abstract available. PMID 31857029
- [Background] Jimenez Diaz VA, Lozano I, Baz Alonso JA, Calvo Iglesias F, Iniguez Romo A. HALT After TAVR: Searching the Bases, Finding the Cusp. JACC Cardiovasc Interv. 2019 May 13;12(9):894-895. doi: 10.1016/j.jcin.2019.02.011. No abstract available. PMID 31072513
- [Background] Jimenez Diaz VA, Tello-Montoliu A, Moreno R, Cruz Gonzalez I, Iniguez Romo A. Reply: The REAC-TAVI Trial: Better Antiplatelet Therapy, Less Haze on the Horizon. JACC Cardiovasc Interv. 2019 Apr 22;12(8):803-804. doi: 10.1016/j.jcin.2019.02.038. No abstract available. PMID 31000022
- [Background] Jimenez Diaz VA, Baz Alonso JA, Estevez Ojea O, Serantes Combo A, Rodriguez Paz CM, Iniguez Romo A. Real-Time Detection of an Acute Cerebral Thrombotic Occlusion During a Transcatheter Valve Intervention. JACC Cardiovasc Interv. 2018 Jul 9;11(13):e103-e104. doi: 10.1016/j.jcin.2018.03.048. Epub 2018 Jun 13. No abstract available. PMID 29908965
- [Background] Kim WK, Pellegrini C, Ludwig S, Mollmann H, Leuschner F, Makkar R, Leick J, Amat-Santos IJ, Dorr O, Breitbart P, Jimenez Diaz VA, Dabrowski M, Rudolph T, Avanzas P, Kaur J, Toggweiler S, Kerber S, Ranosch P, Regazzoli D, Frank D, Landes U, Webb J, Barbanti M, Purita P, Pilgrim T, Liska B, Tabata N, Rheude T, Seiffert M, Eckel C, Allali A, Valvo R, Yoon SH, Werner N, Nef H, Choi YH, Hamm CW, Sinning JM. Feasibility of Coronary Access in Patients With Acute Coronary Syndrome and Previous TAVR. JACC Cardiovasc Interv. 2021 Jul 26;14(14):1578-1590. doi: 10.1016/j.jcin.2021.05.007. PMID 34294400
- [Background] Brouwer J, Nijenhuis VJ, Delewi R, Hermanides RS, Holvoet W, Dubois CLF, Frambach P, De Bruyne B, van Houwelingen GK, Van Der Heyden JAS, Tousek P, van der Kley F, Buysschaert I, Schotborgh CE, Ferdinande B, van der Harst P, Roosen J, Peper J, Thielen FWF, Veenstra L, Chan Pin Yin DRPP, Swaans MJ, Rensing BJWM, van 't Hof AWJ, Timmers L, Kelder JC, Stella PR, Baan J, Ten Berg JM. Aspirin with or without Clopidogrel after Transcatheter Aortic-Valve Implantation. N Engl J Med. 2020 Oct 8;383(15):1447-1457. doi: 10.1056/NEJMoa2017815. Epub 2020 Aug 30. PMID 32865376
- [Result] Jimenez Diaz VA, Tello-Montoliu A, Moreno R, Cruz Gonzalez I, Baz Alonso JA, Romaguera R, Molina Navarro E, Juan Salvadores P, Paredes Galan E, De Miguel Castro A, Bastos Fernandez G, Ortiz Saez A, Fernandez Barbeira S, Raposeiras Roubin S, Ocampo Miguez J, Serra Penaranda A, Valdes Chavarri M, Cequier Fillat A, Calvo Iglesias F, Iniguez Romo A. Assessment of Platelet REACtivity After Transcatheter Aortic Valve Replacement: The REAC-TAVI Trial. JACC Cardiovasc Interv. 2019 Jan 14;12(1):22-32. doi: 10.1016/j.jcin.2018.10.005. PMID 30621974
- [Result] Trejo-Velasco B, Cruz-Gonzalez I, Tello-Montoliu A, Baz-Alonso JA, Salvadores PJ, Moreno R, Romaguera R, Molina-Navarro E, Paredes-Galan E, De-Miguel-Castro A, Bastos-Fernandez G, Ortiz-Saez A, Fernandez-Barbeira S, Iniguez-Romo A, Jimenez-Diaz VA. Influence of Valve Type and Antiplatelet Regimen on Platelet Reactivity After TAVI: Subanalysis of the REAC-TAVI Trial. J Invasive Cardiol. 2020 Dec;32(12):446-452. doi: 10.25270/jic/20.00167. Epub 2020 Aug 10. PMID 32771996
- [Result] Trejo-Velasco B, Tello-Montoliu A, Cruz-Gonzalez I, Moreno R, Baz-Alonso JA, Salvadores PJ, Romaguera R, Molina-Navarro E, Paredes-Galan E, Fernandez-Barbeira S, Ortiz-Saez A, Bastos-Fernandez G, De Miguel-Castro A, Figueiras-Guzman A, Iniguez-Romo A, Jimenez-Diaz VA. Impact of Comorbidities and Antiplatelet Regimen on Platelet Reactivity Levels in Patients Undergoing Transcatheter Aortic Valve Implantation. J Cardiovasc Pharmacol. 2021 Sep 1;78(3):463-473. doi: 10.1097/FJC.0000000000001075. PMID 34117181